CLINICAL TRIAL: NCT01807286
Title: A Phase I/II Clinical Trial of Pomalidomide With Melphalan and Dexamethasone in Patients With Newly Diagnosed Untreated Systemic AL Amyloidosis: Trial Stopped During Phase I
Brief Title: Pomalidomide With Melphalan and Dexamethasone for Untreated Systemic AL Amyloidosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor requested termination
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0215; NCI-2013-02276 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Myeloma
Keywords: Myeloma; Untreated Systemic AL Amyloidosis; Amyloid light-chain (AL) amyloidosis; Pomalidomide; Melphalan; Alkeran; Dexamethasone; Decadron; Questionnaires; Surveys
MeSH Terms: conditions — Neoplasms, Plasma Cell; Amyloidosis | interventions — pomalidomide; Melphalan; Dexamethasone; Calcium Dobesilate; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomalidomide + Melphalan + Dexamethasone (Experimental): Starting dose of Pomalidomide 1 mg/day by mouth on days 1-21. Melphalan 9 mg/m2 by mouth on days 1-4 of every 28-day cycle. Dexamethasone 40 mg/day by mouth on days 1-4. Questionnaires completed at different time points during study.
  Interventions: Drug: Pomalidomide; Drug: Melphalan; Drug: Dexamethasone; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Pomalidomide — Phase I: Starting dose of Pomalidomide 1 mg/day by mouth on days 1-21 of a 28 day cycle.
  Phase II: Starting dose of Pomalidomide maximum tolerated dose from Phase I.
Drug: Melphalan — Phase I and II: 9 mg/m2 by mouth on days 1-4 of a 28-day cycle.
  Other Names: Alkeran
Drug: Dexamethasone — Phase I and II: 40 mg/day by mouth on days 1-4 of a 28 day cycle.
  Other Names: Decadron
Behavioral: Questionnaires — Questionnaires about the feeling in hands and quality of life completed at different time points during the study.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of pomalidomide that can be given in combination with melphalan and dexamethasone that can be given to patients with AL amyloidosis. The safety of this drug combination will also be studied.

Pomalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. This may decrease the growth of cancer cells.

Melphalan is designed to damage the DNA (genetic material) of cells, which may cause cancer cells to die.

Dexamethasone is a corticosteroid that is similar to a natural hormone made by your body. Dexamethasone is often given to Multiple Myeloma (MM) patients in combination with other chemotherapy to treat cancer.

Planned Phase I/II Study terminated early during Phase I portion without continuation to Phase II.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of pomalidomide, based on when you join this study. Up to 4 dose levels of pomalidomide will be tested for the Phase I portion of this study. Up to 30 participants will be enrolled at each dose level in the Phase I portion, and up to 24 participants will be enrolled in Phase II. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of pomalidomide is found.

If you are enrolled in the Phase II portion, you will receive pomalidomide at the highest dose that was tolerated in the Phase I portion.

All participants will receive the same dose level of dexamethasone and melphalan. If intolerable side effects are seen at the lowest dose level, then the melphalan dose will be lowered.

After 2 cycles of therapy, you may be referred to a transplant specialist, if you are eligible for a stem cell transplant.

Study Drug Administration:

Each cycle is 28 days.

Treatment Phase:

You will take pomalidomide pills by mouth on Days 1-21 of each cycle. You should take each dose of pomalidomide at about the same time every day. Swallow the pomalidomide capsules whole with water at the same time each day. Pomalidomide should be taken without food (at least 2 hours before or 2 hours after a meal). Do not break, chew, or open the capsules. If you miss a dose of pomalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (DO NOT take double your regular dose to make up for the missed dose). You should tell the study doctor and/or nurse right away about any missed doses of pomalidomide. If you take more than the prescribed dose of pomalidomide, you should seek emergency medical care, if needed, and contact the study staff right away. You will need to return any unused pomalidomide and empty bottles to the clinic at each study visit.

You will also be given a study drug diary. Each time you take pomalidomide, melphalan or dexamethasone at home, you should write down the date, time, and how many capsules or tablets you took. You should bring the diary in with you at each study visit for the study doctor to review.

On Days 1-4 of each cycle, you will take melphalan pills by mouth one time each day. You should take melphalan in the morning at least 2 hours before or after a meal.

You will take dexamethasone pills on Days 1-4 of each cycle.

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks. You will receive a blood thinner to prevent blood clots. The study doctor will decide what type of blood thinner you will receive.

Maintenance Phase:

You will take pomalidomide pills by mouth on Days 1-28 of each cycle during the maintenance phase. You should take each dose of pomalidomide at about the same time every day. Swallow the pomalidomide capsules whole with water, at the same time each day. Do not break, chew, or open the capsules. If you miss a dose of pomalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (DO NOT take double your regular dose to make up for the missed dose). You should tell the study doctor and/or nurse right away about any missed doses of pomalidomide. If you take more than the prescribed dose of pomalidomide, you should seek emergency medical care, if needed, and contact the study staff right away. You will need to return any unused pomalidomide and empty bottles to the clinic at each study visit.

You will also be given a study drug diary. Each time you take pomalidomide, melphalan, or dexamethasone at home, you should write down the date, time, and how many capsules or tablets you took. You should bring the diary in with you at each study visit for the study doctor to review.

Study Visits:

At every visit you will be asked if you have had any side effects and to list any drugs you may be taking.

Treatment Phase:

On Day 1 of Cycle 1:

* Your medical history will be reviewed and recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be given the study drug diary.
* You will complete 2 questionnaires about quality-of-life, your general health, your level of pain, and how the disease affects you. It will take about 15 minutes to complete the questionnaires.
* Blood (about 1 tablespoon) and urine and/or feces (over 24 hours) will be collected to check the status of the disease.
* Blood (about 1 tablespoon) will be drawn for routine tests. If you are able to become pregnant, a pregnancy test will also be performed.
* If your doctor thinks it is needed, you will have an EKG and an ECHO.

On Days 8 and 22 of Cycle 1:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* If you are able to become pregnant, blood (about 2 teaspoons) will be drawn for a pregnancy test.

On Day 15 of Cycle 1:

* Your medical history will be reviewed and recorded.
* You will have a physical exam including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If you are able to become pregnant, blood (about 2 teaspoons) will be drawn for a pregnancy test.

On Day 1 of Cycles 2 and beyond:

* Your medical history will be reviewed and recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will complete 2 questionnaires about quality-of-life, your general health, your level of pain, and how the disease affects you. It will take about 15 minutes to complete the questionnaires.

I-f your doctor thinks it is needed, blood (about 1 tablespoon) and urine (over 24 hours) will be collected to check the status of the disease.

* Blood (about 1 tablespoon) will be drawn for routine tests. If you are able to become pregnant, a pregnancy test will also be performed.
* Urine will be collected for routine tests.
* If your doctor thinks it is needed, you will have a bone marrow aspiration and biopsy to check the status of your disease and for genetic testing.
* If your doctor thinks it is needed, you will have an EKG and an ECHO.

On Day 15 of Cycles 2 and beyond:

* You will complete a questionnaire about your general health, your level of pain, and how the disease affects you. It will take about 8 minutes to complete the questionnaire.
* If you are able to become pregnant, blood (about 2 teaspoons) will be drawn for a pregnancy test.

Maintenance Phase:

On Day 1 of Cycle 1:

* Your medical history will be reviewed and recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will complete 2 questionnaires about quality-of-life, your general health, your level of pain, and how the disease affects you. It will take about 15 minutes to complete the questionnaires.
* If your doctor thinks it is needed,blood (about 1 tablespoon) and urine (over 24 hours) will be collected to check the status of the disease.
* Blood (about 1 tablespoon) will be drawn for genetic testing.
* Blood (about 1 tablespoon) will be drawn for routine tests. If you are able to become pregnant, a pregnancy test will also be performed.
* Urine will be collected for routine tests.
* If your doctor thinks it is needed, you will have an EKG and an ECHO.

On Day 1 of Cycles 2 and beyond:

* Your medical history will be reviewed and recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will complete 2 questionnaires about quality-of-life, your general health, your level of pain, and how the disease affects you. It will take about 15 minutes to complete the questionnaires.
* If your doctor thinks it is needed, blood (about 1 tablespoon) and urine (over 24 hours) will be collected to check the status of the disease.
* Blood (about 1 tablespoon) will be drawn for routine tests. If you are able to become pregnant, a pregnancy test will also be performed.
* Urine will be collected for routine tests.
* If your doctor thinks it is needed, you will have an EKG and an ECHO.

On Day 15 of Cycles 1 and beyond:

-If you are able to become pregnant, blood (about 2 teaspoons) will be drawn for a pregnancy test.

Length of Study:

The Treatment Phase of the study will take about 6 months to complete. If the study doctor thinks you are benefiting from the study drug combination, you will go into the Maintenance Phase. You can continue taking the study drug(s) until you experience intolerable side effects, the disease gets worse, or the study doctor thinks it is in your best interests to stop.

End-of-Treatment Visit:

If you go off study for any reason, you will have an end-of-treatment visit within 30 days after the last dose of the study drug combination and the following tests and procedures will be performed:

* Your medical history will be reviewed and recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* You will have an ECHO.
* Your performance status will be recorded.
* You will complete 2 questionnaires about quality-of-life, your general health, your level of pain, and how the disease affects you. It will take about 15 minutes to complete the questionnaires.
* Blood (about 1 tablespoon) will be drawn to check the status of the disease.
* Blood (about 1 tablespoon) will be drawn for routine tests. If you are able to become pregnant, a pregnancy test will also be performed 28 days after your last dose of pomalidomide if you have regular periods or 14 and 28 days after your last dose of pomalidomide if you have irregular periods.
* If your doctor thinks it is necessary, you will have a MRI or a CT scan to check the status of the disease.
* If the doctor thinks it is possible, you will have a bone marrow aspiration and biopsy to check the status of disease and for genetic testing.

Long Term Follow-Up:

After the end-of-treatment visit, you will be contacted either by telephone or during one of your standard of care office visits every 3 to 6 months and asked how you are doing. If you are contacted by phone, the call will take about 5 minutes.

This is an investigational study. Pomalidomide, Melphalan, and Dexamethasone are FDA approved and commercially available for the treatment of MM. The study drug combination is not FDA approved or commercially available as a first-line treatment for AL amyloidosis. It is currently being used for research purposes only.

Up to 54 patients will be enrolled at The University of Texas (UT) MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years old.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2; Karnofsky >/= 60%
3. Patients must be willing and able to provide voluntary written informed consent, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care
4. Histologic diagnosis of amyloidosis by Congo red staining of tissue biopsy within 12 months of enrollment.
5. Demonstrable clonal plasma cell disorder based on the presence of an M protein in the serum and/or urine by immunofixation and/or serum free light chain assay, and/or a clonal population of plasma cells in the bone marrow based on kappa/lambda staining of a marrow biopsy.
6. If no demonstrable associated light chain abnormality, then no-light chain amyloidosis should be excluded by checking for transthyretin, fibrinogen A alpha, Amyloid A^3.
7. Patients must have measurable disease, as defined by at least one of the following: Serum or urine immunofixation showing a monoclonal protein and clonal marrow plasmacytosis by marrow biopsy immunohistochemical staining; Free light chains with an abnormal free light chain ratio
8. Symptomatic end organ involvement with amyloidosis as defined previously and to include any one of the following: Renal - albuminuria higher than 0.5 g/day in 24-hour urine analysis; Cardiac - presence of a mean left ventricular wall thickness on echocardiogram more than 11 mm in the absence of a history of hypertension or valvular heart disease, or unexplained low voltage (<0.5 mV) on electrocardiogram; Hepatic - hepatomegaly on physical examination with an alkaline phosphatase level higher than 200 U/L; Gastrointestinal - gastrointestinal amyloid deposits confirmed by tissue biopsy.; Soft-tissue or lymphatic involvement - ascertained based on classic physical exam findings (macroglossia, shoulder pad sign, raccoon eyes, carpal tunnel syndrome, synovial enlargement, firm enlarged lymph nodes) or biopsy.
9. Inclusion Criteria #8 cont... - Nerve - positive history of autonomic or peripheral neuropathy and/or nerve conduction defect documented by electromyogram (EMG)/nerve conduction velocity (NCV) testing.; Skin- measurable skin lesions that are biopsy proven to be amyloidosis
10. No prior therapy for the monoclonal plasma cell disease.
11. Patients must have evidence of adequate bone marrow reserves, as defined by the following pretreatment clinical laboratory values within 14 days of study initiation: Platelet count >/= 100 x 10^9/L without platelet transfusions within 2 weeks of the initiation of treatment; Hemoglobin >/= 8 g/dLwithout red blood cell transfusions within 2 weeks of the initiation of treatment; Absolute neutrophil count (ANC) >/= 1.0x10^9/L without growth factor requirement within 1 week of the initiation of treatment
12. Patients must have evidence of adequate hepatic function, as defined by the following: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 2.5 times the upper limit of normal; Total bilirubin </= 1.5 times the upper limit of normal
13. Patients must have evidence of adequate renal function, as defined by the following: Serum creatinine within the institutional normal limits, OR, if the creatinine is elevated: Creatinine clearance (CrCl) >/= 30 mL/min., as measured by a 24-hour urine collection, or estimated by the Cockcroft and Gault formula: Female CrCl = (140 - age in years) x weight in kg x 0.85/ 72 x serum creatinine in mg/dL ; Male CrCl = (140 - age in years) x weight in kg x 1.00/72 x serum creatinine in mg/dL
14. Patients must have evidence of adequate cardiac function, as defined by the following: Absence of New York Heart Association (NYHA) class III or IV congestive heart failure; Absence of uncontrolled angina or hypertension; Absence of myocardial infarction in the previous 6 months; Absence of clinically significant bradycardia, or other uncontrolled cardiac arrhythmia defined as grade 3 or 4 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0
15. Patients who have undergone any recent major surgery must have done so at least 4 weeks prior to starting therapy with PMD, with the following exceptions:Vertebroplasty and/or kyphoplasty, which must have been performed at least 1 week prior to starting PMD; Planned elective surgery unrelated to the patient's diagnosis of multiple myeloma, such as hernia repair, may be allowed, at the discretion of the principle investigator, as long as it was performed at least 2 weeks prior to starting PMD, and patients have recovered fully from this procedure
16. Male patients must agree to use an adequate method of contraception for the duration of the study since the effects of PMD on the developing human fetus are unknown. If a female partner of a male subject taking Pomalidomide becomes pregnant, the male subject taking Pomalidomide should notify the Investigator immediately. The pregnant female partner should notify their healthcare provider. Female patients must be either post menopausal, free from menses for >/= 2 years, surgically sterilized, or willing to use two adequate barrier methods of contraception to prevent pregnancy, or must agree to abstain from heterosexual activity throughout the study. Female patients of childbearing potential must have a negative serum pregnancy test (Beta-HCG) before receiving the first dose of PMD. The female participant must also follow pregnancy testing requirements as outlined in the POMALYST REMS program.
17. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
18. All study participants must be registered into the mandatory POMALYST REMSTM program, and be willing and able to comply with the requirements of the POMALYST REMSTM program.

Exclusion Criteria:

1. Patients who are receiving any concurrent investigational agent with known or suspected activity against amyloidosis
2. Peripheral neuropathy Grade 2 or higher, as defined by National Cancer Institute Common Terminology Criteria (NCI CTC) version 4.
3. Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure uncontrolled angina, or clinically significant pericardial disease.
4. Stage III cardiac amyloidosis with NT-proBNP> 8000 ng/L.
5. Amyloid-specific syndrome, such as carpal tunnel syndrome or skin purpura as the only evidence of disease. The finding of vascular amyloid only in a bone marrow biopsy specimen or in a plasmacytoma is not indicative of systemic amyloidosis.
6. Presence of non-AL amyloidosis
7. Clinically overt multiple myeloma with definite lytic bone lesions.
8. Other malignancy within the past 5 years. Exceptions include basal cell or non-metastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or FIGO Stage 1 carcinoma of the cervix, or breast or prostate cancer that have been stable on hormonal therapy for at least three years.
9. Concurrent medical condition or disease, such as active systemic infection, uncontrolled diabetes, or pulmonary disease, that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
10. Use of any investigational drugs within 30 days before initiation of study treatment
11. Human immunodeficiency virus (HIV) positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pomalidomide. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
12. Patients with active hepatitis B and/or hepatitis C infection
13. Known hypersensitivity to thalidomide or lenalidomide.
14. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, pomalidomide or similar drugs.
15. Any prior use of thalidomide, lenalidomide or pomalidomide.
16. Known positive for HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Pomalidomide with Melphalan and Dexamethasone (PMD). | 28 days
  Maximum tolerated dose defined as highest dose level at which less than 33% of patients experienced dose-limiting toxicities. Dose-limiting toxicities defined as (grade 4 neutropenia lasting more than 7 days despite G-CSF administration, any other grade 4 hematologic toxicity, any grade 3 non-hematologic toxicity, or a new cycle delay beyond a maximum of 4 weeks) in less than 33% of patients during the first cycle of therapy.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | Response evaluated after a minimum of 2 cycles and a maximum of 6 cycles of 28-day treatment
  CR Rate is number of participants with CR out of total study participants. Complete response defined using treatment response in primary systemic amyloidosis from the 10th International Symposium on Amyloid and Amyloidosis where CR: Serum and urine negative for a monoclonal protein by immunofixation; free light chain ratio normal; marrow <5% plasma cells.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Orlowski, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org